CLINICAL TRIAL: NCT06273098
Title: Understanding and Enhancing Schoolchildren's Bathroom Habits: Uncovering Barriers and Promoting Healthy Bladder Habits
Brief Title: School-Based Bladder Health Intervention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The record was submitted too early. We will need to finalize funding and measured outcomes.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kathleen Kan, Clinical Assistant Professor, Urology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 73162
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Urinary Dysfunction; Lower Urinary Tract Symptoms; Urinary Tract Infections; Urinary Tract Infections in Children
Keywords: School-Based Intervention; Bathroom Policy; Healthy Bladder Behaviors; Bladder Health Education
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Tract Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bladder Health Education (Experimental): Participants in this arm will receive the intervention
  Interventions: Behavioral: Bladder Health Education
- No Bladder Health Education (No Intervention): Participants in this arm will not receive the intervention

INTERVENTIONS:
Behavioral: Bladder Health Education — This will be a combination of bladder health education and awareness events, additional resources such as a water station to support healthy bladder behaviors, and tailored changes to classroom bathroom policies that are TBD (e.g. mobile technology bathroom passes).
  Arms: Bladder Health Education

SUMMARY:
The aim of this study is to promote healthy bladder behaviors among school children. We hypothesize that a combination of bladder health education and awareness events, additional resources such as a water station to support healthy bladder behaviors, and tailored changes to classroom bathroom policies can promote healthy bladder behaviors among school children.

DETAILED DESCRIPTION:
In order to promote healthy bladder behaviors among school children, we will conduct a randomized control trial in schools. The research team will provide support for a combination of bladder health education and awareness events, additional resources such as a water station to support healthy bladder behaviors, and tailored changes to classroom bathroom policies that are TBD (e.g. mobile technology bathroom passes).

The study will involve 4-8 fourth grade classrooms within 2 elementary schools that meet the historical criteria for >50% students receiving free school lunch.

ELIGIBILITY:
Inclusion Criteria:

* 4th grade students from elementary schools that meet the historical criteria for >50% students receiving free school lunch.

Exclusion Criteria:

* Not meet the inclusion criteria

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2028-01-01 (Estimated); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Bathroom use | 4 years
  Individual child's bathroom use (# of bathroom trips measured using mobile technology bathroom passes)
Symptom score | 4 years
  Changes in a child's symptom score (survey questions before, during and after the study)
Urine volume | 4 years
  Changes in a child's volume of urine (child will void into private bathroom before and during the study to understand if their bladder are too full, no direct observation)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Kan, Principal Investigator — Stanford University
Locations (1):
- Stanford Hospital and Clinics, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
Identifiers might be removed from identifiable private information and, after such removal, the information could be used for future research studies or distributed to another investigator for future research studies. Any shared data will be de-identified.